CLINICAL TRIAL: NCT00134407
Title: Postoperative Enteral Feeding or Early Oral Intake at Will. Effects on Clinical Outcome
Brief Title: Postoperative Oral Intake Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NFR 147339/320
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2011-09-05 (Estimated); Status verified 2011-09

CONDITIONS: Postoperative Care
Keywords: Nutrition; Postoperative; oral; jejunal; feeding; Surgery; major; abdominal; adult

INTERVENTIONS:
Procedure: Normal diet
Procedure: Nutrition via jejunal needle-catheter

SUMMARY:
Complete fasting until resumed bowel function after upper abdominal surgery is not beneficial. Enteral feeding has been claimed to be the preferred way of delivering nutritional support postoperatively. Increasing evidence suggests that letting patients eat ("voluntary oral feeding" or "oral intake at will") from the day after the operation is safe. No prospective randomised trial has been undertaken to compare these two regimens. In this study, the investigators will randomise 444 patients, subject to major upper abdominal surgery, into receiving either continuous enteral feeding by needle catheter jejunostomy until resumed bowel function, or to oral intake at will from postoperative day 1. The main endpoints are the incidence rate of major complications and death, as well as a Quality of Life assessment.

Null-Hypothesis:

Routine postoperative feeding by needle catheter jejunostomy after major, upper abdominal surgery has no clinically relevant advantages over early oral intake at will.

DETAILED DESCRIPTION:
Complete fasting until resumed bowel function after upper abdominal surgery is not beneficial. Enteral feeding has been claimed to be the preferred way of delivering nutritional support postoperatively. Increasing evidence suggests that letting patients eat ("voluntary oral feeding" or "oral intake at will") from the day after the operation is safe. No prospective randomised trial has been undertaken to compare these two regimens. In this study, we will randomise 444 patients, subject to major upper abdominal surgery, into receiving either continuous enteral feeding by needle catheter jejunostomy until resumed bowel function, or to oral intake at will from postoperative day 1. The main endpoints are the incidence rate of major complications and death, as well as a Quality of Life assessment.

Null-Hypothesis:

Routine postoperative feeding by needle catheter jejunostomy after major, upper abdominal surgery has no clinically relevant advantages over early oral intake at will.

ELIGIBILITY:
Inclusion Criteria:

* Adults subject to major, upper, open abdominal surgery (exceeding simple cholecystectomies and fundoplications)

Exclusion Criteria:

* Crohns disease
* Mentally disabled
* Pre-op dependency on intravenous (IV) nutrition
* Expected life duration of less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450
Dates: Start 2001-02; Study Completion 2006-06

PRIMARY OUTCOMES:
Major complications within 8 weeks postoperatively

SECONDARY OUTCOMES:
Minor complications
Quality of Life
Use of analgesics
Post-laparotomy bowel movement

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Revhaug, Professor, Study Chair — University of Northern Norway
Locations (1):
- University Hospital Northern Norway,, Tromsø, Tromsø, Norway